CLINICAL TRIAL: NCT05988021
Title: An Open-Label, Phase 1 Study in Healthy Volunteers to Evaluate the Pharmacokinetic Food Effect and Cardiac Safety of CCX168
Brief Title: A Study in Healthy Volunteers to Evaluate the Pharmacokinetic Food Effect and Cardiac Safety of CCX168
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CL007_168
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Anti-neutrophil Cytoplasmic Antibody-associated Vasculitis
Keywords: Vasculitis; Complement; C5aR; Vascular diseases; Cardiovascular diseases; Systemic vasculitis; ANCA
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis; Vascular Diseases; Cardiovascular Diseases; Systemic Vasculitis | interventions — avacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Sequence ABCD (Experimental): Participants assigned to sequence ABCD will receive the following treatments:
  Period 1: Single dose of 30 mg CCX168 after a high-fat, high-calorie meal (Treatment A).
  Period 2: After a washout period of ≥ 10 days, single dose of 30 mg CCX168 in the fasted state (Treatment B).
  Period 3: After a washout period of ≥ 10 days, single dose of 3 mg CCX168 in the fasted state (Treatment C).
  Period 4: 24 hours after the 3 mg CCX168 dose in Period 3, single dose of 100 mg CCX168 on Day 1, and then 100 mg CCX168 twice daily from Day 2 through Day 6. On Day 7, only a morning dose of 100 mg CCX168 (Treatment D).
  Interventions: Drug: CCX168
- Cohort 2: Sequence BACD (Experimental): Participants assigned to sequence BACD will receive the following treatments:
  Period 1: Single dose of 30 mg CCX168 in the fasted state (Treatment B).
  Period 2: After a washout period of ≥ 10 days, single dose of 30 mg CCX168 after a high-fat, high-calorie meal (Treatment A).
  Period 3: After a washout period of ≥ 10 days, single dose of 3 mg CCX168 in the fasted state (Treatment C).
  Period 4: 24 hours after the 3 mg CCX168 dose in Period 3, single dose of 100 mg CCX168 on Day 1, and then 100 mg CCX168 twice daily from Day 2 through Day 6. On Day 7, only a morning dose of 100 mg CCX168 (Treatment D).
  Interventions: Drug: CCX168

INTERVENTIONS:
Drug: CCX168 — Administered orally.

SUMMARY:
The primary objective of this clinical trial is to evaluate the effect of a high-fat, high-calorie meal on the pharmacokinetic (PK) profile of CCX168, following oral administration of a single dose of 30 mg CCX168 to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged 18-55 years inclusive, who are in generally good health, whose body mass index is 19.0 to 32.0 kg/m^2 inclusive;
* Willing and able to give written Informed Consent and to comply with the requirements of the study protocol;
* Negative result of the human immunodeficiency virus screen, the hepatitis B screen, and the hepatitis C screen;
* Judged to be healthy by the Investigator, based on medical history, physical examination (including ECG, and clinical laboratory assessments. Participants with clinical laboratory values that are outside of normal limits and/or with other abnormal clinical findings that are judged by the Investigator not to be of clinical significance may be entered into the study;
* Female participants of childbearing potential, or male participants with partners of childbearing potential may participate if adequate contraception is used during, and for at least 90 days after, any administration of study medication.

Exclusion Criteria:

* Women who are pregnant, lactating, or have a positive serum pregnancy test at screening or check-in (Day -2);
* Myocardial infarction or active ischemic heart disease within 12 months before screening;
* Significant abnormal ECG: Pacemaker, any conduction abnormality associated with a QRS ≥120 msec, poorly-defined or abnormal T wave morphology precluding end of T measurement, abnormal rhythm for age, evidence of previous myocardial infarction (Q waves, S-T segment changes), sinus pauses > 2.5 seconds, ventricular couplets, triplets or other arrhythmia, symptomatic or asymptomatic;
* Has any of the following abnormalities:

  1. Heart rate <40 or >100 bpm
  2. PR interval <110 or ≥220 msec
  3. QRS duration ≥120 msec
  4. QTcF interval <350 or >450 msec;
* History of additional significant risk factors for torsade de pointes, including heart failure, hypokalemia, hypocalcemia, hypomagnesemia, family history of long QT syndrome;
* Used a prescription and/or over-the-counter medication, with the exception of ibuprofen, hormonal contraceptives, and multi-vitamins, within 14 days prior to check-in;
* History within the three months prior to check-in of use of tobacco and/or nicotine-containing products;
* History within one year prior to check-in of illicit drug use;
* History of alcohol abuse at any time in the past;
* Has a history or presence of any form of cancer within the 5 years prior to check-in, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis;
* For at least 14 days prior to check-in and throughout the blood sample collection period, participants will not be allowed to eat any food or drink any beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens) and charbroiled meats;
* History or presence of unexplained syncope or family history of sudden death, or any medical condition or disease which, in the opinion of the Investigator, may place the participants at unacceptable risk for study participation;
* Donated or lost more than 350 mL of blood or blood products within 56 days prior to screening, or donated plasma within 7 days of dosing;
* Participant's hemoglobin less than 11.5 g/dL for women or less than 13.0 g/dL for men at screening or check-in, confirmed by a repeat measurement;
* Participated in any clinical study of an investigational product within 30 days prior to dosing, or within 5 half-lives after dosing;
* Participant has any evidence of hepatic disease; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or bilirubin greater than 1.5 times the upper limit of normal at screening or check-in;
* Participant's white blood cell count is below the lower limit of normal at screening or check-in, confirmed by a repeat measurement;
* Participant has any evidence of renal impairment; serum creatinine greater than 1.5 times the upper limit of normal at screening or check-in;
* Participant's urine tested positive at screening and/or on check-in for any of the following: opioids, amphetamines and methamphetamines, cannabinoids, benzodiazepines, barbiturates, cocaine, cotinine, ecstasy, methadone, phencyclidine, tri-cyclic antidepressants, or alcohol (Breathalyzer test allowed for alcohol).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CCX168 | Up to 35 days
Time of Cmax (Tmax) of CCX168 | Up to 35 days
Area Under the Plasma Concentration-time Curve (AUC) of CCX168 From Time 0 to Time t (AUC0-t) | Up to 35 days
AUC of CCX168 From Time 0 to Infinity (AUC0-inf) | Up to 35 days

SECONDARY OUTCOMES:
Number of Participants Experiencing Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to 35 days
Number of Participants Experiencing Adverse Events (AEs) | Up to 35 days
Number of Participants Experiencing Clinically Significant Changes in Laboratory Parameters | Up to 35 days
Number of Participants Experiencing Clinically Significant Changes in Vital Sign Parameters | Up to 35 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com